CLINICAL TRIAL: NCT05782699
Title: Detection of Impending Reflex Syncope by Means of an Integrated Multisensor Patch-type Recorder
Brief Title: Detecting Syncope by an Integrated Multisensor Patch-type Recorder
Acronym: Patch-VD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Michele Brignole, Principal Investigator, Istituto Auxologico Italiano
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09C126
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Syncope, Vasovagal
Keywords: syncope; tilt table test; blood pressure monitoring
MeSH Terms: conditions — Syncope, Vasovagal; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patch monitoring (Experimental)
  Interventions: Device: BP monitoring during tilt testing
- standard BP monitoring (Active Comparator)
  Interventions: Device: BP monitoring during tilt testing

INTERVENTIONS:
Device: BP monitoring during tilt testing — BP measure at various times during tilt testing

SUMMARY:
The main purpose of this study is to assess the reliability of a new cuffless patch BP monitor in detecting episodes of hypotensive (pre)syncope during tilt testing.

DETAILED DESCRIPTION:
Background While ECG monitoring is a reliable and established method that allows to document bradycardia in a substantial proportion of patients affected by cardioinhibitory reflex syncope, the documentation of a transient hypotension is only seldom achieved in patients affected by hypotensive syncope. Conventional ambulatory blood pressure (BP) monitoring (ABPM) has important limitations due to the short period of monitoring (usually 24-48 hours) and the intermittent nature of BP measurements (usually every 15-20 min).

The main purpose of this study is to assess the reliability of a new cuffless patch BP monitor in detecting episodes of hypotensive (pre)syncope. Secondary aim regards the estimation of feasibility of this tool.

Method The study is a prospective intrapatient comparison between BP measured by mean of a cuffless patch BP monitor (RootiRX System, Rooti Labs Ltd., Taipei, Taiwan) and by mean of the standard method during tilt testing.

Study design BP values observed during tilt testing baseline and at the time of impeding syncope will be measured by mean of the RootiRX device and will be compared with the standard of reference. BP will be recorded at rest at baseline, shortly after upright in tilting position (at stabilization), at the time of occurrence of syncope (presyncope) or, alternatively at the time of maximum hypotensive effect, if syncope will not occur, and finally in the recovery period at the end of the test after returning in supine position.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients,
* >18 years of age,
* referred for tilt testing because affected by suspected reflex syncope

Exclusion Criteria:

* Incapability to perform tilt testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
BP pattern | 2 hours
  Difference between baseline (rest) BP and BP at the (pre)syncopal event ("Delta BP slope") during tilt testing with RootiRx and with standard method

SECONDARY OUTCOMES:
BP drop | 2 hours
  Absolute BP values during tilt event with RootiRx and with Finometer

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: Upon reasonable request after the publication of the principal study
Access Criteria: m.brignole@auxologico.it